CLINICAL TRIAL: NCT04503200
Title: Double Guidewire Technique Versus Transpancreatic Precut in Patients With Repetitive Unintentional Cannulation of the Pancreatic Duct.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hany Shehab, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DGWRCT
Record Dates: First submitted 2020-08-04; First posted 2020-08-07 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Endoscopic Retrograde Cholangiopancreatography; Common Bile Duct Diseases; Transpancreatic Precut; Precut; Double Guidewire
MeSH Terms: conditions — Common Bile Duct Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Double guidewire (Active Comparator)
  Interventions: Procedure: Double guidewire
- Transpancreatic precut (Active Comparator)
  Interventions: Procedure: Transpancreatic precut

INTERVENTIONS:
Procedure: Double guidewire — After the 3rd passage of the guidewire into the pancreatic duct, the catheter will be removed leaving the guidewire in place. The catheter will be re-inserted and a second guidewire will be used and directed above the pancreatic wire in the 11-12 o'clock direction to attempt cannulation of the common bile duct.
  Arms: Double guidewire
Procedure: Transpancreatic precut — After the 3rd passage of the guidewire unintentionally into the pancreatic duct, the guidewire will be left in the pancreatic duct, a sphincterotome will be used to cut in the direction of 11-12 o'clock attempting to deroof the pancreatic duct and gain access into the common bile duct. The wire will then be retracted and reinserted in the direction of the cut to attempt cannulation of the common bile duct.
  Arms: Transpancreatic precut

SUMMARY:
Difficult cannulation of the common bile duct is encountered in about 10%of ERCP procedures. This frequently happens in the form of repeated unintentional cannulation of the pancreatic duct. Two valid options are available to facilitate cannulation at this point: Double guidewire technique or performing a transpancreatic precut. This is a randomized trial comparing the efficacy and Safety of double guidwire technique versus transpancreatic precut after three unintentional passages of the guidewire into the pancreatic duct.

ELIGIBILITY:
Inclusion Criteria:

* unintentional cannulation of the pancreatic duct 3 times
* Consenting to join the study

Exclusion Criteria:

* Previous ERCP with or without previous sphincterotomy
* Known coagulopathy

  * - Pregnancy
  * - Known acute pancreatitis at the time of procedure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-08-15 (Estimated); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Cannulation success | Within 10 minutes
  Proportion of patients with successful cannulation of the common bile duct
Rate of post-ERCP pancreatitis | up to 24 hours after the procedure
  Proportion of patients suffering post-ERCP pancreatitis

SECONDARY OUTCOMES:
Time to successful cannulation | Within 10 minutes
  Time to achieve cannulation after the 3rd passage of the guidewire into the pancreatic duct

CONTACTS AND LOCATIONS:
Overall Officials: Hany M Shehab, Study Chair — Kasr-Elaini Faculty of Medicine
Locations (1):
- Cairo University, Cairo, Egypt